CLINICAL TRIAL: NCT04962841
Title: Cognitive and Physical Impairment in Frail Older Adults
Brief Title: Nutraceuticals and Drug Treatment in Frail Older Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Pasquale Mone, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: Campania Nord
Record Dates: First submitted 2021-07-10; First posted 2021-07-15 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Frailty
Keywords: frailty; cognitive impairment; physical impairment; older adults
MeSH Terms: conditions — Frailty; Cognitive Dysfunction | interventions — Dietary Supplements; Nebivolol; Sertraline; Rivastigmine; Metformin; Ramipril; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail older adults treated with nutraceuticals and drugs
  Interventions: Other: Nutraceuticals
- Frail older adults not treated with nutraceuticals and drugs

INTERVENTIONS:
Other: Nutraceuticals — To observe the effect on cognitive and physical impairment.
  Other Names: empaglifozin; nebivolol; sertraline; rivastigmine; metformin; ramipril; amlodipine
  Groups: Frail older adults treated with nutraceuticals and drugs

SUMMARY:
Frailty is a multidimensional condition due to reserve loss leading to physical and cognitive impairment that is very common in older adults; in fact, its incidence increases with age. Frail older adults present a high risk of adverse events such as disability, hospitalization and mortality. It is very important to check comorbidities and complications to reduce the incidence of cognitive and physical impairment.

DETAILED DESCRIPTION:
Frailty is a multidimensional condition due to reserve loss leading to physical and cognitive impairment that is very common in older adults; in fact, its incidence increases with age. Frail older adults present a high-risk of adverse events such as disability, hospitalization and mortality. It is very important to check comorbidities and complications to reduce the incidence of cognitive and physical impairment; hence, clinical evaluation is the main goal to get an early diagnosis and a timely treatment for cognitive impairment. Considering this background, the study will investigate the effects of nutraceuticals and drug treatment on cognitive impairment in frail older adults. In this scenario, global cognitive function will be evaluated with Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) test and physical impairment with the Fried criteria and 5-metres gait speed test.

ELIGIBILITY:
Inclusion Criteria:

* age > 65 years;
* a frailty status.

Exclusion Criteria:

* age < 65 years.
* no frailty status.
* left ventricular ejection fraction <25%, with previous myocardial infarction or previous PPCI or/and coronary by-pass grafting.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Frail older adults.
Sampling Method: Probability Sample
Enrollment: 485 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | July 2021
  Global cognitive impairment

SECONDARY OUTCOMES:
5 metres gait speed test | July 2021
  Physical impairment

OTHER OUTCOMES:
Correlation between MMSE/MoCA and 5 metres gait speed test | July 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Pasquale Mone, Naples, It, Italy

REFERENCES:
- [Background] Cortes-Canteli M, Iadecola C. Alzheimer's Disease and Vascular Aging: JACC Focus Seminar. J Am Coll Cardiol. 2020 Mar 3;75(8):942-951. doi: 10.1016/j.jacc.2019.10.062. PMID 32130930
- [Background] Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, Popma JJ, Ferrucci L, Forman DE. Frailty assessment in the cardiovascular care of older adults. J Am Coll Cardiol. 2014 Mar 4;63(8):747-62. doi: 10.1016/j.jacc.2013.09.070. Epub 2013 Nov 27. PMID 24291279
- [Background] Jung HW, Baek JY, Jang IY, Guralnik JM, Rockwood K, Lee E, Kim DH. Short Physical Performance Battery as a Crosswalk Between Frailty Phenotype and Deficit Accumulation Frailty Index. J Gerontol A Biol Sci Med Sci. 2021 Nov 15;76(12):2249-2255. doi: 10.1093/gerona/glab087. PMID 33780526
- [Derived] Mone P, Pansini A, Jankauskas SS, Varzideh F, Kansakar U, Lombardi A, Trimarco V, Frullone S, Santulli G. L-Arginine Improves Cognitive Impairment in Hypertensive Frail Older Adults. Front Cardiovasc Med. 2022 Apr 12;9:868521. doi: 10.3389/fcvm.2022.868521. eCollection 2022. PMID 35498050
- [Derived] Mone P, Lombardi A, Gambardella J, Pansini A, Macina G, Morgante M, Frullone S, Santulli G. Empagliflozin Improves Cognitive Impairment in Frail Older Adults With Type 2 Diabetes and Heart Failure With Preserved Ejection Fraction. Diabetes Care. 2022 May 1;45(5):1247-1251. doi: 10.2337/dc21-2434. PMID 35287171